CLINICAL TRIAL: NCT02983305
Title: Optical Head-Mounted Display Technology for Low Vision Rehabilitation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Joshua Ehrlich, Professor, University of Michigan
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HUM00110408
Record Dates: First submitted 2016-11-04; First posted 2016-12-06 (Estimated); Results first posted 2019-10-09 (Actual); Last update posted 2019-10-09 (Actual); Status verified 2019-09

CONDITIONS: Retinal Dystrophies; Healthy
MeSH Terms: conditions — Retinal Dystrophies | interventions — Smart Glasses

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Retinal Dystrophy (Experimental): Subjects with retinal dystrophy will have their visual field, gait and self-reported mobility tested at baseline. Subjects will then be fit with a head-mounted display and undergo a brief training with the investigators to learn about use of the device. After a 2 week period of in-home adaptation to the device, their visual field, gait and self-reported mobility will be retested.
  Interventions: Device: Head-Mounted Display
- Healthy Age-Matched Controls (Experimental): Age-matched control subjects without eye disease will have their visual field, gait and self-reported mobility tested at baseline. Control subjects will then be fit with a head-mounted display and undergo a brief training with the investigators to learn about use of the device. After a 2 week period of in-home adaptation to the device, their visual field, gait and self-reported mobility will be retested.
  Interventions: Device: Head-Mounted Display

INTERVENTIONS:
Device: Head-Mounted Display — Head-mounted displays (HMD) are a class of technology that are worn on the user's head and project an image either in front of or into the eye.
  Other Names: Epson Moverio

SUMMARY:
The goal of this study is to examine the ability of optical head-mounted display technology to enlarge the visual field of patients with severe visual field loss due to retinal dystrophy and to improve mobility and patient-reported outcomes.

DETAILED DESCRIPTION:
Worldwide it is estimated that 191 million people have moderate to severe visual impairment (MSVI) and an additional 32.4 million are blind. Patients with uncorrectable MSVI may undergo low vision rehabilitation (LVR), which has been shown to improve functional abilities, such as mobility. However, existing LVR strategies do not adequately address severe visual field constriction.

In this pilot study, the investigators will test the hypothesis that optical head-mounted display (HMD) technology expands constricted visual fields and improves mobility outcomes for patients with retinal dystrophy. We will use the Moverio HMD platform which is considered a non-significant risk device. Outcomes for patients with retinal dystrophy will be compared to normal age-matched controls.

ELIGIBILITY:
Inclusion criteria for subjects with retinal dystrophy:

* diagnosis of retinal dystrophy
* severe vision loss that constitutes legal blindness
* able to perform a reliable Goldmann visual field test
* constricted visual field less than or equal to 20 degrees by Goldmann perimetry using the III4e stimulus in at least one eye with best-corrected visual acuity ≥ 20/60

Inclusion criteria for control subjects:

* healthy controls
* visit history with the Comprehensive and Pediatric Ophthalmology Services at the University of Michigan
* able to perform a reliable Goldmann visual field test

Exclusion criteria for subjects with retinal dystrophy:

* movement disorder that precludes evaluation of mobility
* functional vision loss
* pregnant women

Exclusion criteria for control subjects:

* visually significant ocular condition other than correctable refractive error
* movement disorder that precludes evaluation of mobility
* functional vision loss
* pregnant women

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2017-06-26 (Actual); Primary Completion 2018-11-21 (Actual); Study Completion 2018-11-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joshua R Ehrlich, MD, MPH, Principal Investigator — University of Michigan
Locations (1):
- Kellogg Eye Center, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Retinal Dystrophy | Healthy Age-Matched Controls
Started | 12 | 10
Completed (Participants were deemed to have not completed the study if they contributed incomplete data.) | 10 | 10
Not Completed | 2 | 0
Not completed — incomplete data | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Retinal Dystrophy | Healthy Age-Matched Controls | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 33.5 [23 to 37] | 33 [23.5 to 39.75] | 33.5 [23 to 39.5]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 5 | 10
  Male | 5 | 5 | 10
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Visual Field Area [Median (Inter-Quartile Range); unit: degrees^2] — Average of both eyes visual fields at baseline (no intervention).
  degrees^2 | 568.96 [232.40 to 742.94] | 19280.09 [18441.30 to 19388.97] | 19009.42 [12235.76 to 19355.28]
Gait Speed [Median (Inter-Quartile Range); unit: meters per second] — Average of both feet at baseline (no intervention).
  meters per second | 1.27 [1.10 to 1.31] | 1.25 [1.21 to 1.42] | 1.26 [1.15 to 1.32]

OUTCOME MEASURES:

1. Primary Outcome: Change in the Planimetric Area of Goldmann Visual Field With the Use of Head-mounted Display Technology Compared to Baseline (Measured in Degrees Squared)
Description: Using computer software we will calculate the area of participants' Goldmann visual fields in order to obtain a summary quantitative measurement of the extent of peripheral vision.
  Average of both eyes visual fields with intervention.
Time Frame: Baseline and two to four weeks
Measure: Median (Inter-Quartile Range); unit: degrees^2
Arm/Group | Retinal Dystrophy | Healthy Age-Matched Controls
Number analyzed (Participants) | 10 | 10
degrees^2 | 563.08 [331.97 to 715.60] | -3799.19 [-4482.99 to -2598.07]
Statistical Analysis 1: Comparison: Retinal Dystrophy vs Healthy Age-Matched Controls; Test of equivalence of visual field area at baseline; Test type: Equivalence — Mann-Whitney U test was used to test equivalence of this outcome measure for the two study arms at baseline; p = .0001, Wilcoxon (Mann-Whitney) — P < .05 was considered a priori to be statistically significant
Statistical Analysis 2: Comparison: Retinal Dystrophy vs Healthy Age-Matched Controls; Test of equivalence of visual field area under intervention conditions; Test type: Equivalence — Mann-Whitney U test was used to test equivalence of this outcome measure for the two study arms under intervention conditions; p = 0.0001, Wilcoxon (Mann-Whitney) — P < .05 was considered a priori to be statistically significant
Statistical Analysis 3: Comparison: Retinal Dystrophy vs Healthy Age-Matched Controls; Comparison between study arms of the change in the visual field area (average of both eyes) detected between baseline and intervention; Test type: Equivalence — Mann-Whitney U test was used to test non-equivalence of this outcome measure for the two study arms under intervention conditions; p = .003, Wilcoxon (Mann-Whitney) — P < .05 was considered a priori to be statistically significant

2. Secondary Outcome: Change in Gait Speed Compared to Baseline (Measured in Seconds)
Description: Gait speed will be measured using an inertial measurement unit attached to participants' shoes and will quantify the time taken to move from the beginning to end of a short mobility course.
  Average of data from both feet with intervention.
Time Frame: Baseline and two to four weeks
Measure: Median (Inter-Quartile Range); unit: meters per second
Arm/Group | Retinal Dystrophy | Healthy Age-Matched Controls
Number analyzed (Participants) | 10 | 10
meters per second | -.01 [-.05 to 0.00] | -.01 [-.05 to .05]
Statistical Analysis 1: Comparison: Retinal Dystrophy vs Healthy Age-Matched Controls; Test of equivalence of gait speed at baseline; Test type: Equivalence — Mann-Whitney U test was used to test equivalence of this outcome measure for the two study arms at baseline; p = 0.38, Wilcoxon (Mann-Whitney) — P < .05 was considered a priori to be statistically significant
Statistical Analysis 2: Comparison: Retinal Dystrophy vs Healthy Age-Matched Controls; Test of equivalence of gait speed under intervention conditions; Test type: Equivalence — [test comment as in outcome 1, analysis 2]; p = 0.27, Wilcoxon (Mann-Whitney) — P < .05 was considered a priori to be statistically significant
Statistical Analysis 3: Comparison: Retinal Dystrophy vs Healthy Age-Matched Controls; Comparison between study arms of the change in the gait speed detected between baseline and intervention; Test type: Equivalence — [test comment as in outcome 1, analysis 3]; p = 0.79, Wilcoxon (Mann-Whitney) — P < .05 was considered a priori to be statistically significant

ADVERSE EVENTS:
Time Frame: Through study completion, an average of 2-4 weeks.
Arm/Group | Retinal Dystrophy | Healthy Age-Matched Controls
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/10
Other Adverse Events (participants affected / at risk) | 0/12 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-06-15): https://cdn.clinicaltrials.gov/large-docs/05/NCT02983305/Prot_SAP_000.pdf